CLINICAL TRIAL: NCT03163433
Title: Feedback in the Consultation - a Dialogue-based Tool in Personalised Care Planning Using Systematic Patient Involvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Cancer Society (Other); AmbuFlex (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Feedback in the consultation
Record Dates: First submitted 2017-05-08; First posted 2017-05-23 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Melanoma; Quality of Life
Keywords: Patient activation measure; Self-efficacy; Patient participation in research; Patient reported outcome measures
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: The intervention takes place at a highly specialized university hospital i Denmark. Two other higly specialized Danish hospitals recruit patients for the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback in the consultation (Experimental): Feedback in the consultation is the intervention. Patients complete PROM before each consultation and take part in a dialogue about the results with their physician.
  Interventions: Behavioral: Feedback in the consultation
- Control (No Intervention): Usual consultations

INTERVENTIONS:
Behavioral: Feedback in the consultation — Patients will complete electronic Patient Reported Outcome Measures (PROM) before the consultation at the hospital. The results are fed back to physicians. In the consultation patients will systematically participate in a dialogue with their physician about issues that are most important for the patients.
  Arms: Feedback in the consultation

SUMMARY:
The aim of the study is to examine the potentials of involving patients with metastatic melanoma in their own care planning through systematic use of patient-reported outcome measures (PROM). Furthermore, to examine the outcome of health-related quality of life, self-efficacy and impact on the patient-physician interaction.

Patients (N=282) will be included from three highly specialized hospitals in Denmark. At one hospital patients will complete PROM before each consultation during a year (intervention group). At the two other hospitals patients will not complete PROM (control group). In addition to baseline, measurements will take place after three, six and 12 months. The project is organized and executed with patient involvement in the research process.

DETAILED DESCRIPTION:
Background:

In recent years, treatment of metastatic melanoma has changed significantly, which has led to improved prognosis and greater expectations for the future. However, new concerns in relation to health-related quality of life and coping with disease in everyday life have emerged. Patient-reported outcome measures (PROM) is a promising tool to strengthen patient involvement. By systematically reporting real time PROM to the physician prior to a consultation, it may generate a continuous feedback loop, by which the patient physician dialogue can focus on what is most important to the patient.

Hypothesis:

The aim of the study is to investigate the potentials of using PROM as a dialogue-based tool. We hypothesize that PROM as a dialogue-based tool can:

* Improve patients' knowledge, skills, and confidence for managing their health and healthcare
* Reduce the perceived burden of physical symptoms and emotional dysfunction
* Improve the quality of the patient-physician interaction

Material and methods:

In this prospective study patients (N=282) will be included from three highly specialized hospitals in Denmark. At Aarhus University Hospital, patients will complete electronic PROM before the consultation and systematically participate in a dialogue about their self-assessments for a duration of one year (intervention group). At Herlev Hospital and Odense University Hospital, patients will not complete PROM (control group). In addition to baseline, self-reported measurements will take place after three, six and 12 months.

To address the patient perspective, patients with melanoma are involved in the project management. A steering group with scientists and patient representatives has been established. This group have chosen the relevant PROM, determined primary objectives and given feedback on the written information material for the intervention by looking at relevance and readability. Moreover the group will ensure optimal implementation if results are promising. In addition, a patient focus group will be established to discuss how PROM should be used in the consultation and how patient involvement is expressed in practice. The recruitment of patients to these groups will be made in cooperation with the association for patients with melanoma and clinical practice where the patients are treated.

Perspectives If results are positive, the intervention will be easy to apply to routine settings and in a slightly adjusted form in other groups of cancer patients too.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving treatment for metastatic melanoma in Denmark
* Manage to read and speak Danish

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Patient Activation Measure (PAM) | 1 year
  A 13-item measurement of patients' knowledge, skills, and confidence for managing their health and healthcare

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy - Melanoma (FACT-M) | 1 year
  A 51-item measurement of quality of life
Cancer Behavior Inventory (CBI) | 1 year
  A 14-item measurement of self-efficacy in patients with cancer
Perceived Efficacy in Patient-Physician Interaction (PEPPI) | 1 year
  A 5-item measurement of patient-physician interaction

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Lomborg, Professor, Study Chair — University of Aarhus
Locations (1):
- Aarhus University Hospital, Department of Oncology, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skovlund PC, Nielsen BK, Thaysen HV, Schmidt H, Finset A, Hansen KA, Lomborg K. The impact of patient involvement in research: a case study of the planning, conduct and dissemination of a clinical, controlled trial. Res Involv Engagem. 2020 Jul 19;6:43. doi: 10.1186/s40900-020-00214-5. eCollection 2020. PMID 32699648